CLINICAL TRIAL: NCT06261125
Title: Efficacy and Safety of Stereotactic Body Radiotherapy Followed by Adebrelimab and Lenvatinib for Hepatocellular Carcinoma With Abdominal Lymph Node Metastases: A Two-arm, Phase II Trial
Brief Title: Combination of SBRT, PD-L1 Inhibitor, and Lenvatinib in Hepatocellular Carcinoma (HSBRT2401)
Acronym: HSBRT2401
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mian XI (Other)
Responsible Party: Sponsor-Investigator, Mian XI, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2023-718
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Radiotherapy; Immunotherapy; Targeted therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): This arm includes the patients who previously had not received PD-1/PD-L1 antibody. Patients assigned to this arm will receive SBRT followed by adebrelimab and lenvatinib. The prescribed dose of SBRT is 33-48 Gy in 6 fractions over 2 weeks. Then all patients will receive lenvatinib (12 mg/day for bodyweight ≥60 kg or 8 mg/day for bodyweight <60 kg) orally once daily in combination with adebrelimab 1200 mg every 3 weeks for up to 35 cycles. The first course of adebrelimab will be given within 1 week after completion of SBRT.
  Interventions: Radiation: Stereotactic body radiotherapy; Drug: Adebrelimab; Drug: Lenvatinib
- Arm B (Experimental): This arm includes the patients who had progressed after receiving PD-1/PD-L1 antibody. Patients assigned to this arm will receive SBRT followed by adebrelimab and lenvatinib. The prescribed dose of SBRT is 33-48 Gy in 6 fractions over 2 weeks. Then all patients will receive lenvatinib (12 mg/day for bodyweight ≥60 kg or 8 mg/day for bodyweight <60 kg) orally once daily in combination with adebrelimab 1200 mg every 3 weeks for up to 35 cycles. The first course of adebrelimab will be given within 1 week after completion of SBRT.
  Interventions: Radiation: Stereotactic body radiotherapy; Drug: Adebrelimab; Drug: Lenvatinib

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Patients in both cohorts will receive stereotactic body radiotherapy (SBRT) using volumetric arc therapy. The prescribed dose is 33-48 Gy in 6 fractions over 2 weeks.
  Other Names: SBRT
Drug: Adebrelimab — All patients will reveive adebrelimab 1200 mg every 3 weeks for up to 35 cycles after the completion of SBRT.
  Other Names: SHR-1316
Drug: Lenvatinib — All patients will receive lenvatinib (12 mg/day for bodyweight ≥60 kg or 8 mg/day for bodyweight <60 kg) orally once daily after the completion of SBRT.
  Other Names: Lenvima

SUMMARY:
Abdominal lymph node metastasis (LNM) is one of the major modes of extrahepatic metastasis in hepatocellular carcinoma (HCC). Immunotherapy targeting the PD-1/PD-L1 checkpoints combined with targeted therapy is the standard treatment for HCC with abdominal LNM, but the outcome remains very poor, with an objective response rate of 5% to 30%. Previous studies have demonstrated that stereotactic body radiotherapy (SBRT) is an effective local treatment for HCC with abdominal LNM, with a high response rate of 60% to 80%. However, intrahepatic dissemination and distant metastasis remains the major recurrence pattern after SBRT in these patients, suggesting radiotherapy should be combined with systematic treatment. Recently, the combination of immunotherapy with SBRT has shown promising activity in HCC. The aim of this study was to investigate the efficacy and safety of SBRT followed by adebrelimab (an anti-PD-L1 antibody) and lenvatinib in HCC patients with portal abdominal LNM.

DETAILED DESCRIPTION:
A total of 60 HCC patients (2 cohorts) with abdominal LNM will be enrolled to receive SBRT followed by adebrelimab (an anti-PD-L1 antibody) and lenvatinib. Arm A included the patients who previously had not received PD-1/PD-L1 antibody, and Arm B included the patients who had progressed after receiving PD-1/PD-L1 antibody.

Patients in both cohorts will receive stereotactic body radiotherapy (SBRT) using volumetric arc therapy. The prescribed dose is 33-48 Gy in 6 fractions over 2 weeks. Then all patients will receive lenvatinib (12 mg/day for bodyweight ≥60 kg or 8 mg/day for bodyweight <60 kg) orally once daily in combination with adebrelimab 1200 mg every 3 weeks for up to 35 cycles. The first course of adebrelimab will be given within 1 week after completion of SBRT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed hepatocellular carcinoma or diagnosed by American Association for the Study of Liver Disease criteria;
2. Presence of abdominal metastatic lymph nodes confirmed by CT or MRI, the sum of the maximum diameter of lymph nodes ≤10 cm, and at least one of which is measurable according to the RECIST 1.1 Criteria;
3. Previous local treatment for intrahepatic lesion and systemic anti-tumor therapy are allowed; no matter whether the disease progressed or not;
4. Less than 3 active intrahepatic lesions with a total diameter of less than 10 cm; Portal vein invasion is allowed; absence of other extrahepatic metastasis disease except abdominal LNM;
5. Cohort 1: Patients who never received PD-1/PD-L1 antibody therapy; Cohort 2: patients who had tumor progression after previous PD-1/PD-L1 antibody therapy.
6. Age at diagnosis 18 to 75 years;
7. Eastern Cooperative Oncology Group performance status ≤ 2
8. Child-Pugh class A liver function;
9. Normal liver volume greater than 700 ml;
10. Estimated life expectancy ≥12 weeks;
11. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥ 3.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L; b. platelets ≥ 50×109/L; c. hemoglobin ≥ 9g/dL; d. serum albumin ≥ 2.8g/dL; e. total bilirubin ≤ 1.5×ULN, ALT, AST and/or AKP ≤ 2.5×ULN; f. serum creatinine ≤ 1.5×ULN or creatinine clearance rate >60 mL/min;
12. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Diffuse hepatocellular carcinoma;
2. Patients who have previously been treated with lenvatinib or PD-1/PD-L1 antibody but could not be tolerated;
3. Patients with other extrahepatic metastasis disease except abdominal LNM;
4. A history of abdominal radiotherapy;
5. Known or suspected allergy or hypersensitivity to monoclonal antibodies;
6. Patients who have a preexisting or coexisting bleeding disorder;
7. Female patients who are pregnant or lactating;
8. Inability to provide informed consent due to psychological, familial, social and other factors;
9. A history of malignancies other than hepatocellular carcinoma before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer;
10. A history of diabetes for more than 10 years and poorly controlled blood glucose levels;
11. Patients who cannot tolerate radiotherapy due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia;
12. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
13. A history of interstitial lung disease or non-infectious pneumonia;
14. A history of active pulmonary tuberculosis infection within 1 year or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal anti-tuberculosis treatment;
15. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C (positive for hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay);
16. Any unstable situation that may endanger the safety and compliance of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From date of enrollment until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 36 months.
  Three-year follow-up from the date of enrollment to the date of disease progression or last follow-up

SECONDARY OUTCOMES:
Overall survival (OS) | From date of enrollment until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 36 months.
  Three-year follow-up from the enrollment to the date of death from any cause or date of lost follow-up
Overall response rate (ORR) | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  Tumor response was evaluated every 9 weeks after the completion of radiotherapy based on CT or MRI scan.
Disease control rate (DCR) | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  The proportion of patients with complete response, partial response, or stable disease according to RECIST criteria.
Duration of response (DOR) | From date of first CR/PR to the date of first PD according to RECIST criteria, assessed up to 36 months.
  From the date of first CR/PR to the date of first PD.
Treatment-related adverse events | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  Incidence of treatment-related adverse events as assessed by CTCAE v4.0.

OTHER OUTCOMES:
Correlation between serum cytokines and overall survival and immune-related adverse events | From date of enrollment to the date of last follow-up, assessed up to 36 months.
  The correlation between dynamic change of serum cytokines (IL-2R, IL-6, IL-13, IL-8, CCL3, CD40, and CD274) during treatment and survival outcomes and immune-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mian Xi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Mian Xi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Result] Wang Y, Li Q, Zhang L, Liu S, Zhu J, Yang Y, Liu M, Zhang Y, Xi M. Efficacy and Dose-Response Relationship of Stereotactic Body Radiotherapy for Abdominal Lymph Node Metastases from Hepatocellular Carcinoma. Oncologist. 2023 Jun 2;28(6):e369-e378. doi: 10.1093/oncolo/oyad083. PMID 37011232
- [Result] Kim HJ, Park S, Kim KJ, Seong J. Clinical significance of soluble programmed cell death ligand-1 (sPD-L1) in hepatocellular carcinoma patients treated with radiotherapy. Radiother Oncol. 2018 Oct;129(1):130-135. doi: 10.1016/j.radonc.2017.11.027. Epub 2018 Jan 30. PMID 29366520
- [Result] Chiang CL, Chiu KWH, Chan KSK, Lee FAS, Li JCB, Wan CWS, Dai WC, Lam TC, Chen W, Wong NSM, Cheung ALY, Lee VWY, Lau VWH, El Helali A, Man K, Kong FMS, Lo CM, Chan AC. Sequential transarterial chemoembolisation and stereotactic body radiotherapy followed by immunotherapy as conversion therapy for patients with locally advanced, unresectable hepatocellular carcinoma (START-FIT): a single-arm, phase 2 trial. Lancet Gastroenterol Hepatol. 2023 Feb;8(2):169-178. doi: 10.1016/S2468-1253(22)00339-9. Epub 2022 Dec 15. PMID 36529152
- [Result] Finn RS, Ikeda M, Zhu AX, Sung MW, Baron AD, Kudo M, Okusaka T, Kobayashi M, Kumada H, Kaneko S, Pracht M, Mamontov K, Meyer T, Kubota T, Dutcus CE, Saito K, Siegel AB, Dubrovsky L, Mody K, Llovet JM. Phase Ib Study of Lenvatinib Plus Pembrolizumab in Patients With Unresectable Hepatocellular Carcinoma. J Clin Oncol. 2020 Sep 10;38(26):2960-2970. doi: 10.1200/JCO.20.00808. Epub 2020 Jul 27. PMID 32716739